CLINICAL TRIAL: NCT05738603
Title: The Hypotension Prediction Index in Free Flap Transplant in Head and Neck Surgery - a Prospective Randomized Controlled Trial.
Brief Title: The Hypotension Prediction Index in Free Flap Transplant in Head and Neck Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Szrama (Other)
Responsible Party: Sponsor-Investigator, Jakub Szrama, Principal Investigator, Poznan University of Medical Sciences
Organization: Poznan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 560/22
Record Dates: First submitted 2023-01-15; First posted 2023-02-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hypotension; Head and Neck Cancer; Perioperative Complication; Postoperative Complications
Keywords: Hypotension; Hypotension Prediction Index; Free Flap Transplant; Head and Neck Cancer; Perioperative Complications
MeSH Terms: conditions — Hypotension; Head and Neck Neoplasms; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: This prospective, randomized, controlled clinical trial will be performed in Poznan University of Medical Science Hospital. Patients fulfilling the inclusion criteria (see below) will be randomly assigned to receive invasive blood pressure monitoring + standard medical therapy (group A) or the hemodynamic monitoring with the Hypotension Prediction Index software (group B).
Who Masked: Participant
Masking Description: The studied patients will be blinded to the enrolled group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Therapy Group (No Intervention): The standard therapy group patients will have invasive blood pressure monitoring + standard medical therapy. The therapeutic decision regarding treatment of hypotension, the use of fluids and vasopressors will be determined by the anaesthesia team. The decisions will be based on the information from the standard invasive blood pressure monitoring.
- Hypotension Prediction Index Group (Experimental): The HPI-group will have the HPI based monitoring with the Acumen IQ sensor (Edwards Lifesciences) and the HPI algorithm connected also to the HemoSphere platform (Edwards Lifesciences). The hemodynamic management will be based on the HPI indications and the specific algorithm, which considers hypovolemia, impaired contractility and vasodilatation. An alert pops up on the monitor screen when the HPI values exceeds 85 and then the clinician needs to make therapeutic decision in order to avoid the hypotensive episode.
  Interventions: Device: Hypotension Prediction Index

INTERVENTIONS:
Device: Hypotension Prediction Index — Hemodynamic perioperative monitoring with the Hypotension Prediction Index
  Arms: Hypotension Prediction Index Group

SUMMARY:
The aim of the current study is to evaluate the effects of the Hypotension Prediction Index (HPI) on the degree of intraoperative hypotension in patients undergoing free flap surgery. The hypothesis is that implementation of the HPI algorithm will reduce the time-weighted average (TWA) intraoperative hypotension below a threshold of 65 mmHg (16), and to reveal the relationship between the episodes of hypotension and free flap viability and function.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualified to head and neck free flap surgery
* Written informed consent

Exclusion Criteria:

* Patients under 18 years
* Lack of health insurance
* Pregnancy
* Known history of congenital heart disease, severe aortic and/or mitral stenosis, heart failure and ejection fraction < 35 %
* Persistent atrial fibrillation and other arrhythmias impairing arterial pressure-based cardiac output (APCO) monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
TWA Mean Arterial Pressure (MAP) < 65 mmHg | From the beginning of the anesthesia to the end of anesthesia
  TWA - MAP < 65 mmHg - time weighed average = (depth of hypotension in millimeters of mercury below a MAP of 65 mmHg x time in minutes spent below MAP of 65mmHg)/total duration of operation in minutes

SECONDARY OUTCOMES:
TWA - MAP < 60 mmHg | From the beginning of the anesthesia to the end of anesthesia
  time weighed average = (depth of hypotension in millimeters of mercury below a MAP of 60 mmHg x time in minutes spent below MAP of 60 mmHg)/total duration of operation in minutes
TWA - MAP < 55 mmHg | From the beginning of the anesthesia to the end of anesthesia
  time weighed average = (depth of hypotension in millimeters of mercury below a MAP of 55 mmHg x time in minutes spent below MAP of 55 mmHg)/total duration of operation in minutes
30 day mortality | 30 days
  30 day mortality
Length of hospitalisation | From date of randomisation to the date of hospital discharge or date of death, whichever came first, assesed up to 3 months
  Length of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Szrama, Ph.D., Principal Investigator — Poznan Univeristy of Medical Sciences, Department of Anesthesiology, Intensive Therapy
Locations (1):
- Department of Anesthesiology, Intensive Therapy and Pain Management, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564
- [Background] Gu WJ, Hou BL, Kwong JSW, Tian X, Qian Y, Cui Y, Hao J, Li JC, Ma ZL, Gu XP. Association between intraoperative hypotension and 30-day mortality, major adverse cardiac events, and acute kidney injury after non-cardiac surgery: A meta-analysis of cohort studies. Int J Cardiol. 2018 May 1;258:68-73. doi: 10.1016/j.ijcard.2018.01.137. Epub 2018 Feb 2. PMID 29429638
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827
- [Background] Maheshwari K, Shimada T, Yang D, Khanna S, Cywinski JB, Irefin SA, Ayad S, Turan A, Ruetzler K, Qiu Y, Saha P, Mascha EJ, Sessler DI. Hypotension Prediction Index for Prevention of Hypotension during Moderate- to High-risk Noncardiac Surgery. Anesthesiology. 2020 Dec 1;133(6):1214-1222. doi: 10.1097/ALN.0000000000003557. PMID 32960954
- [Background] Grundmann CD, Wischermann JM, Fassbender P, Bischoff P, Frey UH. Hemodynamic monitoring with Hypotension Prediction Index versus arterial waveform analysis alone and incidence of perioperative hypotension. Acta Anaesthesiol Scand. 2021 Nov;65(10):1404-1412. doi: 10.1111/aas.13964. Epub 2021 Aug 31. PMID 34322869
- [Derived] Szrama J, Gradys A, Wozniak A, Nowak Z, Bartkowiak T, Lohani A, Zwolinski K, Koszel T, Kusza K. The Hypotension Prediction Index in Free Flap Transplant in Head and Neck Surgery: Protocol of a Prospective Randomized Controlled Trial. Life (Basel). 2025 Mar 4;15(3):400. doi: 10.3390/life15030400. PMID 40141745